CLINICAL TRIAL: NCT00381654
Title: A Phase 1, Sequential Cohort, Dose Escalation Trial to Determine the Safety, Tolerability, and Maximum Tolerated Dose of Daily Oral Administration of AV-412 in Patients With Refractory or Relapsed Solid Tumor Malignancies
Brief Title: Safety/Tolerability Study of AV-412 in Subjects With Refractory or Relapsed Solid Tumor Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study did not meet pre-specified objectives.
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-412-06-101
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-09

CONDITIONS: Tumor
Keywords: Solid Tumors; Tyrosine Kinases
MeSH Terms: conditions — Neoplasms | interventions — MP 412

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Daily oral administration of AV-412
  Interventions: Drug: AV-412

INTERVENTIONS:
Drug: AV-412 — Solid oral dosage; 4 dosage strengths; 25, 50, 100, or 200 mg per capsule Dosing Frequency: Once daily dosing for 4 weeks (4 weeks equals 1 cycle)

SUMMARY:
AV-412 is a new oral therapy developed to inhibit the growth of solid tumors in patients who have not responded to standard therapy or surgical interventions, or who have experienced relapse. This study will test the safety of AV-412 and determine the maximum tolerated dose for the treatment of solid tumors.

DETAILED DESCRIPTION:
Although progress has been made, patients with malignancies often either progress after the traditional approach of chemotherapy, surgery, or radiotherapy, or are not candidates for these approaches because of the advances stage of disease. Novel therapies that may offer greater potential than those currently available are urgently needed.

AV 412 is a potent inhibitor of human epidermal growth factor family receptor tyrosine kinases (TKIs) and represents a growing class of anti-cancer agents. The recent introduction of TKIs has opened the door to new approaches to cancer treatment in which the goals of therapy are to halt disease progression, ameliorate symptoms, and improve patient quality of life. AV412 may inhibit growth of solid tumors, with fewer and less debilitating side effects.

This study is designed to determine the safety, tolerability and maximum tolerated dose of daily oral administration of AV 412. Patients will be assigned to escalating drug dose cohorts to determine the optimal dose. Evaluations to determine tolerability include PK, PD, and the adverse events which occur during the course of study drug administration.

ELIGIBILITY:
Criteria for Inclusion:

1. ≥ 18 year old males or females
2. Documented measurable or evaluable solid tumor malignancy that is relapsed, refractory, locally advanced, or metastatic
3. Patients entered to MTD Cohort B must have:

   * Histologically or cytologically confirmed NSCLC
   * No prior therapy with erlotinib, gefitinib, or any other EGFR-kinase inhibitor
   * Previously documented exon 19 deletion and/or exon 21 L858R mutations
   * Measurable disease according to RECIST
4. Disease that is currently refractory to, or not amenable to, standard therapy
5. Disease that is currently not amenable to surgical intervention, due to either medical contraindications or nonresectability of the tumor
6. Karnofsky performance status ≥ 70%, life expectancy ≥ 3 months
7. No childbearing potential or use of effective contraception by all fertile male and female patients, during the study and for 3 months after the last dose of study drug
8. Ability to give written informed consent

Criteria for Exclusion:

1. Pregnant or lactating women
2. Primary CNS malignancies; active CNS metastases
3. Hematologic malignancies (includes: leukemia, any form; lymphoma; and multiple myeloma)
4. Active second malignancy or history of another malignancy within 2 years with the exception of:

   * Treated, non-melanoma skin cancers
   * Treated CIS of the breast or cervix
   * Controlled, superficial bladder carcinoma
   * T1a or b prostate carcinoma involving < 5% of resected tissue and PSA within normal limits (WNL)
5. Any of the following hematologic abnormalities:

   * Hemoglobin ≤ 9.0 g/dL
   * ANC < 1,500 per mm3
   * Platelet count < 100,000 per mm3
6. Any of the following serum chemistry abnormalities:

   * Total bilirubin > 1.5 × the ULN
   * AST or ALT ≥ 3 × the ULN (≥ 5 × if due to hepatic involvement by tumor)
   * Serum albumin < 2.5 g/dL
   * Creatinine ≥ 1.5 × ULN (or calculated CLCR < 50 mL/min/1.73 m2)
7. Significant cardiovascular disease, including:

   * CHF requiring therapy
   * Ventricular arrhythmia requiring therapy
   * Any conduction disturbance (including patients with QTc interval prolongation > 0.47 sec, history of a severe arrhythmia, or history of a familial arrhythmia [eg, WPW])
   * Angina pectoris requiring therapy
   * LVEF < 50% by MUGA or Echocardiogram
   * Uncontrolled HTN
   * MI within 6 months of study entry
   * NYHA > Class I
8. Significant gastrointestinal abnormalities, including:

   * Requirement for IV alimentation
   * Prior surgical procedures affecting absorption
   * Active peptic ulcer disease
   * ≥Grade 2 diarrhea due to any etiology
9. Known history of significant ophthalmologic abnormalities, including:

   * Severe dry-eye syndrome
   * Keratoconjunctivitis sicca
   * Sjogren's syndrome
   * Severe exposure keratopathy
   * Disorders increasing risk for epithelium-related complications
10. Serious/active infection; infection requiring parenteral antibiotics
11. Inadequate recovery from prior antineoplastic therapy
12. Inadequate recovery from any prior surgical procedure; major surgical procedure within 2 weeks
13. Life-threatening illness or organ system dysfunction compromising safety evaluation
14. Psychiatric disorder, altered mental status precluding informed consent or necessary testing
15. Inability to comply with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, and dose-limiting toxicities (DLT), and determine the maximum tolerated dose (MTD) of AV-412 when administered once daily by the oral route for 4 weeks (4 weeks equals one dosing cycle) | one year

SECONDARY OUTCOMES:
To characterize the pharmacokinetic (PK) profile of AV-412 in all patients. Extensive PK collection and assay to be performed in expanded MTD Cohorts | 18 months
Evaluate potential pharmacodynamic (PD) markers of AV-412 action, in expanded MTD Cohorts ONLY | two years
Preliminary evaluation of the antineoplastic activity of AV-412 (assessed by evidence and duration of disease stabilization or objective response, and time to disease progression) | two years

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, PhD, Principal Investigator — Johns Hopkins University; Justina L Martinez, MD, Principal Investigator — Hospital Universitatrio Austral; Carmen S. Puparelli, MD, Principal Investigator — Instituto Médico Especializado Alexander Fleming; Belén R. Viquiera, M.D., Principal Investigator — Centro Integral Oncológica Clara Campal
Locations (3):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States
- Argentina (2):
  - Hospital Universitatrio Austral, Buenos Aires
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires

REFERENCES:
- See also: Aveo Pharmaceutical, Inc home page — http://aveopharma.com